CLINICAL TRIAL: NCT05993039
Title: Comparison of Inhalational Anesthesia and Total Intravenous Anesthesia on Surgical Field Quality and Post-operative Recovery in Endoscopic Tympanoplasty
Brief Title: Inhalational Anesthesia vs TIVA in Endoscopic Tympanoplasty
Acronym: TIVA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Our Lady of the Lake Hospital (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Leslie Son, Research Scientist-Study Coordinator, Our Lady of the Lake Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIVA in Ear Surgery
Record Dates: First submitted 2023-07-20; First posted 2023-08-15 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Perforated Eardrum
Keywords: tympanoplasty; Inhalational anesthesia; total intravenous anesthesia; intraoperative blood loss
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — Propofol; Remifentanil

STUDY DESIGN:
Intervention Model Description: double-blinded randomized control
Who Masked: Participant, Care Provider
Masking Description: In the operating room, in order to blind the surgeon to the type of anesthesia used, a surgical drape will be placed in between the subject and the anesthesia team to conceal the anesthesia machinery and equipment. A sham intravenous pole will be at the anesthesia workstation for those subjects in the control arm to contribute to the blinding of the surgeon. Patients will not be informed about which arm they are randomly assigned to and only the anesthesiologist will be aware prior to the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhalational Anesthesia (Active Comparator): Adults:
  The control group will receive general inhalational anesthesia (sevoflurane, isoflurane). The will be induced with fentanyl 1-2µg/kg, propofol 2mg/kg, lidocaine 1mg/kg. After orotracheal intubation, anesthesia will be maintained with isoflurane 1.5-2% or sevoflurane 1-2%.
  Children (12 or younger) induced with a combination of volatile anesthetic gases, including sevoflurane (up to 8%) and nitrous oxide gas (up to 70%). Those who are older than 12 will have an intravenous line placed in the preoperative area and as such will be induced with remifentanil and propofol as above. For maintenance, children in the control arm will receive 0.6 - 1.5% sevoflurane.
  Interventions: Drug: Isoflurane Inhalant Product; Drug: Sevoflurane inhalant product
- Total Intravenous Anesthesia (TIVA) (Active Comparator): Adults:
  The comparator arm will receive total intravenous anesthesia (propofol and remifentanil). They will be induced with fentanyl 1-2µg/kg, propofol 2mg/kg, and lidocaine 1mg/kg. After orotracheal intubation, anesthesia will be maintained with propofol 100-200mcg/kg/min, remifentanil 0.05-2µg/kg/min.
  Children (12 or younger) induced with a combination of volatile anesthetic gases, including sevoflurane (up to 8%) and nitrous oxide gas (up to 70%). Those who are older than 12 will have an intravenous line placed in the preoperative area and as such will be induced with remifentanil and propofol as above. For maintenance, they will receive 100-200mcg/min propofol and 0.05-2µg/kg/min remifentanil.
  Interventions: Drug: Propofol injection; Drug: Remifentanil Injection

INTERVENTIONS:
Drug: Isoflurane Inhalant Product — 1.5-2%
  Arms: Inhalational Anesthesia
Drug: Sevoflurane inhalant product — 1-2% adults 0.6-1.5% Children
  Arms: Inhalational Anesthesia
Drug: Propofol injection — 1mg/kg-mcg/kg/min adults 100-200mcg/kg/min children
  Arms: Total Intravenous Anesthesia (TIVA)
Drug: Remifentanil Injection — 0.05-2ug/kg/min adults and children
  Arms: Total Intravenous Anesthesia (TIVA)

SUMMARY:
This study aims to prospectively compare surgical field quality and intraoperative blood loss between general inhalational anesthesia to total intravenous anesthesia (TIVA) alone in subjects undergoing endoscopic ear surgery. A secondary objective is to compare rates of emergence delirium and total recovery time between the two groups.

DETAILED DESCRIPTION:
In sinus surgery, TIVA has been described as a possible advantage in the use of endoscopic ear surgery. However, to date, there are no studies that examine blood loss, surgical field quality, and recovery in TIVA compared to inhalational anesthesia in the setting of endoscopic ear surgery. The hypothesis is that in patients who undergo endoscopic tympanoplasty, those who receive TIVA will have reduced intraoperative blood loss, improved surgical field quality, and reduced emergence agitation than those who receive inhalational anesthesia. This study will be a prospective double-blinded randomized control trial consisting of subjects undergoing endoscopic tympanoplasty surgery to assess intraoperative blood loss, surgical field quality, rates of emergence delirium, and recovery time.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of all ages
* Scheduled to undergo an endoscopic tympanoplasty

Exclusion Criteria:

* Individuals with anticoagulation disorders
* Those receiving anticoagulation therapy currently

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical Field Quality | Post-Operative evaluation (within 2 weeks)
  Neurotologists will evaluate endoscopic video clips from each surgery to assess clarity of field at different points in the surgery using the Boezaart scale grading system. It is a scale from 0-5, with 0 being the most favorable outcome and 5 being the least favorable outcome.
Intra-operative blood loss | 1-2 hours during surgery
  Intraoperative blood loss will be determined by measuring the total number of pledgets needed to attain hemostatsis. This will be a general observation with the more pledgets needed to stop bleeding in the surgical area indicates more possible blood loss than the procedures with that require less pledgets.

SECONDARY OUTCOMES:
Emergent Delirium and Recovery Time-Riker Scale | Immediately After extubation
  Sedation and agitation will be assessed immediately after extubation using the Riker Sedation-Agitation Scale (SAS) which is on scale of 1-7 with 1 being the most favorable (easier to rouse/calm but responsive) and 7 being the least favorable (deeply sedated/higher agitation).
Emergent Delirium and Recovery Time-Richmond Scale | Immediately After extubation
  Sedation and agitation will be assessed immediately after extubation using a second scale known as the Richmond Agitation-Sedation Scale (RASS). The RASS is on a scale of -5 to +4, with higher/more positive scores indicating worse outcomes (aka more aggressive behavior) and lower scores indicating better outcomes (less responsiveness). A score of 0(Zero) indicates a calm but alert patient.
Post-operative pain or complications | 0-1 hour post-operative
  Patients will recover for 1 hour in the post-anesthesia care unit, and a well-trained nurse blinded to the randomized study group will evaluate pain intensity by using the numeric rating scale (0-10 range, with higher scores indicating worse pain) at three intervals: immediately after arrival, 30 minutes after arrival, and 60 minutes after arrival. Any rescue analgesics that are administered will be documented. Patients will be observed postoperatively for any adverse events, as is standard procedure. Any other adverse features such as nausea, vomiting, or changes in vision or color will be followed for 30 days post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Mehta, MD, Principal Investigator — Our Lady of the Lake Hospital
Locations (1):
- Our Lady of the Lake Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No